CLINICAL TRIAL: NCT02916992
Title: Prevalence of Birt-Hogg-Dubé Syndrome Among Patients With (Hereditary) Spontaneous Pneumothorax
Brief Title: Prevalence of Spontaneous Pneumothorax in BHD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hans Smit (Other)
Collaborators: Prof. Dr. Jaap Swieringa stichting (Unknown); Mr. Willem Bakhuys Roozeboomstichting (Unknown); Rijnstate Hospital (Other)
Responsible Party: Sponsor-Investigator, Hans Smit, MD, PhD, Free University Medical Center
Organization: Free University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014-0525; 50605 (Registry Identifier: ABR number); 2014-1386 (Registry Identifier: METc); NL50605.091.14 (Registry Identifier: NL nummer)
Record Dates: First submitted 2016-01-23; First posted 2016-09-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Spontaneous Pneumothorax
Keywords: spontaneous pneumothorax; familial pneumothorax; Birt-Hogg-Dube syndrome; prevalence; FLCN mutation; Lung cysts; BHD; inherited disease; genetic disease; primary pneumothorax; CAT scan; CT scan
MeSH Terms: conditions — Pneumothorax; Birt-Hogg-Dube Syndrome; Cystic Disease Of Lung; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spontaneous pneumothorax patients 1 (Active Comparator): Patients who were treated for spontaneous pneumothorax in Rijnstate hospital. "Interventions": visit to out-patient clinic,CT scan of pulmones.
  Interventions: Radiation: CT scan of the thorax; Genetic: blood sample for FLCN mutation analyses
- Spontaneous pneumothorax patients 2 (Active Comparator): Patients who were treated for spontaneous pneumothorax in Rijnstate hospital. "Interventions": withdrawal of blood sample for DNA analyses,
  Interventions: Radiation: CT scan of the thorax; Genetic: blood sample for FLCN mutation analyses

INTERVENTIONS:
Radiation: CT scan of the thorax — A low dose CT scan of the thorax (2mSv) wil be performed once.
Genetic: blood sample for FLCN mutation analyses — A venous punction in order to withdraw 16ml blood is undertaken once.

SUMMARY:
To assess the prevalence of BHD (Birt-Hogg-Dubé syndrome) among patients with spontaneous pneumothorax. Patients who were treated for primary spontaneous pneumothorax in Rijnstate hospital are to be included. Patients will receive a questionnaire. When given consent, the investigators will invite them for a one-time visit to the out-patient clinic. Patients will be asked for a blood sample to determine pathogenic FLCN (folliculin) mutations and a pulmonary CT scan for evaluation of presence of lung cysts.

DETAILED DESCRIPTION:
Based on the results of the pilot study in VUmc *Free University Medical Center), in which 3 out of 40 tested patients had a pathological FLCN mutation, the investigators decided to extend the study to a second center; Rijnstate Hospital Arnhem. In this hospital a retrospective search was performed; patients who were treated for primary spontaneous pneumothorax were included. In the dossiers the investigators searched for medical history, pneumothorax side and recurrence, diagnostic imaging, treatment, co-morbidity, complications of treatment, skin abnormalities, kidney disease, smoking behavior, medication, and familial incidence of pneumothorax and other diseases. Patients will receive a letter with explanation of the research and a questionnaire in which the investigators ask them their about the medical status, co-morbidity, pneumothorax (number and side), smoking behavior, use of drugs, familial incidence of pneumothorax and other diseases.

The population will be formed out of patients who have returned the fully filled in questionnaire and who have given permission to receive information for further research. This further information will consist of an information letter on BHD syndrome and a consent form for a one-time visit to the out-patient clinic of Rijnstate hospital. Investigators expect that about 200 patients will return the fully filled in questionnaire and give their consent for further research. In a one-time visit in out-patient clinic, there will be given personal information on BHD syndrome and there will be performed physical examination for finding fibrofolliculomas. A pulmonary CT scan for evaluation of presence of lung cysts will be performed. Two samples of venous blood will be collected to access information on DNA diagnostics for pathogenic FLCN mutations. These are associated with the BHD syndrome. This last diagnostic testing will be performed in VUmc (Vrije Universiteit medisch centrum or Free University Medical Centre).

ELIGIBILITY:
Inclusion Criteria:

* treated in Rijnstate hospital for primary spontaneous pneumothorax
* informed consent

Exclusion Criteria:

* secondary or iatrogenic pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
presence of pathogenic FLCN mutations | 6 months
  by assessing blood samples

SECONDARY OUTCOMES:
presence of lung cysts | 6 months
  visible on pulmonary low dose CT

CONTACTS AND LOCATIONS:
Overall Officials: Pieter E. Postmus, MD, PhD, Study Chair — The Clatterbridge Cancer Centre; Hans JM Smit, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johannesma PC, Thunnissen E, Postmus PE. Lung cysts as indicator for Birt-Hogg-Dube syndrome. Lung. 2014 Feb;192(1):215-6. doi: 10.1007/s00408-013-9522-0. Epub 2013 Oct 22. PMID 24146214
- [Background] Toro JR, Wei MH, Glenn GM, Weinreich M, Toure O, Vocke C, Turner M, Choyke P, Merino MJ, Pinto PA, Steinberg SM, Schmidt LS, Linehan WM. BHD mutations, clinical and molecular genetic investigations of Birt-Hogg-Dube syndrome: a new series of 50 families and a review of published reports. J Med Genet. 2008 Jun;45(6):321-31. doi: 10.1136/jmg.2007.054304. Epub 2008 Jan 30. PMID 18234728
- [Background] Houweling AC, Gijezen LM, Jonker MA, van Doorn MB, Oldenburg RA, van Spaendonck-Zwarts KY, Leter EM, van Os TA, van Grieken NC, Jaspars EH, de Jong MM, Bongers EM, Johannesma PC, Postmus PE, van Moorselaar RJ, van Waesberghe JH, Starink TM, van Steensel MA, Gille JJ, Menko FH. Renal cancer and pneumothorax risk in Birt-Hogg-Dube syndrome; an analysis of 115 FLCN mutation carriers from 35 BHD families. Br J Cancer. 2011 Dec 6;105(12):1912-9. doi: 10.1038/bjc.2011.463. PMID 22146830
- [Background] Toro JR, Pautler SE, Stewart L, Glenn GM, Weinreich M, Toure O, Wei MH, Schmidt LS, Davis L, Zbar B, Choyke P, Steinberg SM, Nguyen DM, Linehan WM. Lung cysts, spontaneous pneumothorax, and genetic associations in 89 families with Birt-Hogg-Dube syndrome. Am J Respir Crit Care Med. 2007 May 15;175(10):1044-53. doi: 10.1164/rccm.200610-1483OC. Epub 2007 Feb 22. PMID 17322109
- [Background] Johannesma PC, Reinhard R, Kon Y, Sriram JD, Smit HJ, van Moorselaar RJ, Menko FH, Postmus PE; Amsterdam BHD working group. Prevalence of Birt-Hogg-Dube syndrome in patients with apparently primary spontaneous pneumothorax. Eur Respir J. 2015 Apr;45(4):1191-4. doi: 10.1183/09031936.00196914. Epub 2014 Dec 23. No abstract available. PMID 25537564
- [Background] Johannesma PC, Lammers JW, van Moorselaar RJ, Starink TM, Postmus PE, Menko FH. [Spontaneous pneumothorax as the first manifestation of a hereditary condition with an increased renal cancer risk]. Ned Tijdschr Geneeskd. 2009;153:A581. Dutch. PMID 19857281
- [Background] Ren HZ, Zhu CC, Yang C, Chen SL, Xie J, Hou YY, Xu ZF, Wang DJ, Mu DK, Ma DH, Wang Y, Ye MH, Ye ZR, Chen BF, Wang CG, Lin J, Qiao D, Yi L. Mutation analysis of the FLCN gene in Chinese patients with sporadic and familial isolated primary spontaneous pneumothorax. Clin Genet. 2008 Aug;74(2):178-83. doi: 10.1111/j.1399-0004.2008.01030.x. Epub 2008 May 25. PMID 18505456
- [Background] Warren MB, Torres-Cabala CA, Turner ML, Merino MJ, Matrosova VY, Nickerson ML, Ma W, Linehan WM, Zbar B, Schmidt LS. Expression of Birt-Hogg-Dube gene mRNA in normal and neoplastic human tissues. Mod Pathol. 2004 Aug;17(8):998-1011. doi: 10.1038/modpathol.3800152. PMID 15143337
- [Background] Nickerson ML, Warren MB, Toro JR, Matrosova V, Glenn G, Turner ML, Duray P, Merino M, Choyke P, Pavlovich CP, Sharma N, Walther M, Munroe D, Hill R, Maher E, Greenberg C, Lerman MI, Linehan WM, Zbar B, Schmidt LS. Mutations in a novel gene lead to kidney tumors, lung wall defects, and benign tumors of the hair follicle in patients with the Birt-Hogg-Dube syndrome. Cancer Cell. 2002 Aug;2(2):157-64. doi: 10.1016/s1535-6108(02)00104-6. PMID 12204536
- [Background] Furuya M, Nakatani Y. Birt-Hogg-Dube syndrome: clinicopathological features of the lung. J Clin Pathol. 2013 Mar;66(3):178-86. doi: 10.1136/jclinpath-2012-201200. Epub 2012 Dec 8. PMID 23223565
- [Background] Kilincer A, Ariyurek OM, Karabulut N. Cystic lung disease in birt-hogg-dube syndrome: a case series of three patients. Eurasian J Med. 2014 Jun;46(2):138-41. doi: 10.5152/eajm.2014.31. PMID 25610314
- [Background] Auerbach A, Roberts DH, Gangadharan SP, Kent MS. Birt-Hogg-Dube syndrome in a patient presenting with familial spontaneous pneumothorax. Ann Thorac Surg. 2014 Jul;98(1):325-7. doi: 10.1016/j.athoracsur.2013.09.022. PMID 24996715
- [Derived] Sriram JD, van de Beek I, Johannesma PC, van Werkum MH, van der Wel TJWT, Wessels EM, Gille HJJP, Houweling AC, Postmus PE, Smit HJM. Birt-Hogg-Dube syndrome in apparent primary spontaneous pneumothorax patients; results and recommendations for clinical practice. BMC Pulm Med. 2022 Aug 26;22(1):325. doi: 10.1186/s12890-022-02107-7. PMID 36028846
- Available data/document: Study Protocol: NL50605.091.14 — https://www.toetsingonline.nl/to/ccmo_search.nsf/Searchform?OpenForm — ABR form (Algemeen Beoordelings en Registratie formulier; document of dutch board of human research (Centrale Commissie Mensgebonden Onderzoek)